CLINICAL TRIAL: NCT06222333
Title: Can Breathing Exercise Reduce Pulmonary Complications in Rib Fractures: Randomized Prospective Study
Brief Title: Breathing Exercise for Rib Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, İsmail DAL, Assistant Professor Literally: Doctor Teaching Member, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KastamonuU1
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Rib Fractures; Spirometry
MeSH Terms: conditions — Rib Fractures | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory physiotherapy group (Experimental): In this group of patients, in addition to routine analgesic treatment, triflow use and deep breathing training would be given by the physiotherapist. Patients in this group will do breathing exercises 8 hours a day, 10 times an hour
  Interventions: Behavioral: Respiratory physiotherapy
- Routine treatment group (Active Comparator): Patients in the control group will receive conservative treatment consisting of paracetamol and dexketoprofen.
  Interventions: Drug: Conservative Treatment

INTERVENTIONS:
Behavioral: Respiratory physiotherapy — In this group of patients, in addition to routine analgesic treatment, triflow use and deep breathing training would be given by the physiotherapist. Patients in this group will do breathing exercises 8 hours a day, 10 times an hour.
  Other Names: Triflow
  Arms: Respiratory physiotherapy group
Drug: Conservative Treatment — Patients in the control group will receive conservative treatment consisting of paracetamol and dexketoprofen.
  Other Names: Control
  Arms: Routine treatment group

SUMMARY:
Respiratory physiotherapy is routinely performed after thoracic surgery operations to increase lung expansion and prevent pulmonary complications such as atelectasis and pneumonia. It is a controversial issue whether respiratory physiotherapy reduces pulmonary complications in rib fractures. In our study, patients with rib fractures will be divided into two groups. In the control group, standard treatment consisting of routine analgesic treatments will be applied. In the other group, respiratory physiotherapy will be applied with triflu for 8 hours a day. At the end of the study, pulmonary complications in both groups will be compared.

DETAILED DESCRIPTION:
Patients between the ages of 18 and 100 who will apply to our hospital due to rib fractures between April 2024 and April 2025 will be evaluated. Patients who meet the inclusion criteria will be included in the study. Patients will be divided into two groups using randomization blocks. Patients in the control group will receive conservative treatment consisting of paracetamol and dexketoprofen. In the other group of patients, in addition to conservative treatment, triflow breathing exercise will be applied for 8 hours a day. Respiratory function test pain scores and pulmonary complications of patients in the two groups will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* Isolated thoracic injury within 24 hours
* Age between 18-100

Exclusion Criteria:

* Pneumothorax and hemothorax requiring intervention at admission
* Injury severity index >16
* COPD, Atshma
* Extrathoracic trauma

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
FEV1, FVC, FEV1/FVC results on day 7 | 7 days
  FEV1, FVC, FEV1/FVC

SECONDARY OUTCOMES:
Number of Participants with Pneumonia | 7 days
  Clinical and radiological diagnosis of pneumonia
FEV1, FVC, FEV1/FVC results on day 2 | 2 days
  FEV1, FVC, FEV1/FVC

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Yes
Time Frame: Data will be available permanently on 1.4.2025
Access Criteria: Upon reasonable request principal investigator will share date